CLINICAL TRIAL: NCT00879593
Title: Potential Role for Nocturnal PtcCO2 Monitoring in the Close Follow up of ALS Patients.
Brief Title: Nocturnal PtcCO2 Monitoring in Patients With Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association Nationale pour les Traitements A Domicile, les Innovations et la Recherche (Other)
Responsible Party: Principal Investigator, DELRIEU Jacqueline, PhD, Association Nationale pour les Traitements A Domicile, les Innovations et la Recherche
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ANTADIR PTcCO2/SLA
Record Dates: First submitted 2009-04-09; First posted 2009-04-10 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PtcCO2 (Experimental)
  Interventions: Device: PtcCO2

INTERVENTIONS:
Device: PtcCO2 — Nocturnal assessment will be performed during the initial polysomnography (and at 6 months) with a combined PtcCO2/pulse oxymetry TOSCA500 Radiometer monitoring evaluating different physiological parameters.

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a neurodegenerative disease affecting motoneurons, with a prevalence around 5/100.000. Respiratory muscle involvement is a major feature in ALS and remains the main prognostic factor. Timing and rate of progression of this respiratory muscle involvement is also highly variable among individuals.

Respiratory manifestations justify a careful follow up including clinical evaluation, pulmonary function tests and blood gases. Prognostic value of respiratory muscle assessment has been clearly demonstrated in ALS, although several cut off values have been published. The clinical benefit of non invasive ventilation (NIV) is well established in ALS, but the optimal criteria for its initiation remain debated .

The 1999 consensus for NIV selected classical criteria to consider NIV in patients with respiratory symptoms suggesting hypoventilation: daytime hypercapnia (PaCO2 > 45 mmHg), nocturnal SaO2 < 89 % more than 5 consecutive minutes and for progressive neuromuscular disorders (NMD) (mainly ALS), a vital capacity (VC) < 50 % pred or a PImax < 60 cmH2O.

Besides daytime clinical and PFT assessment, nocturnal evaluation is essential in ALS. The prevalence of sleep apnea ranges from 16 % to 76 %.

Transcutaneous PCO2 (tcPCO2) is an attractive technique to evaluate non invasively nocturnal hypoventilation. The technique is well validated in different settings. Its use in neuromuscular disorders (NMD) is recent. In particular one study has demonstrated a high predictive value of tcPCO2 for the development of daytime hypoventilation within 1 year. To our knowledge, this technique has not been specifically assessed in ALS. There is a potential role for nocturnal PtcCO2 monitoring in the close follow up of ALS patients. Indeed, a close respiratory follow up of ALS patients is essential to determine the optimal timing of NIV, avoiding the occurence of unexpected acute respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Amyotrophic lateral sclerosis :definite, probable or probable with EMG (Airlie House Criteria, 1998).
* Forced vital capacity >70% pred.
* Daytime PaCO2 <43 mmHg.
* Venous HCO3- <28 mmol/L

Exclusion Criteria:

* Patients unable to perform pulmonary function tests or nocturnal recordings.
* Coexisting significant lung disease: moderate to severe asthma or COPD
* Current NIV, CPAP or oxygen therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-04; Primary Completion 2014-06 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Nocturnal Transcutaneous PCO2 | 6 months

SECONDARY OUTCOMES:
Pulmonary function | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thierry PEREZ, MD, Principal Investigator — CHRU LILLE
Locations (2):
- France (2):
  - PEREZ, Lille
  - Pôle des maladies respiratoires et service EFR- Centre hospitalier Regional Universitaire, Lille